CLINICAL TRIAL: NCT03890588
Title: A Technology-Driven Intervention to Improve Identification and Management of Chronic Kidney Disease in Primary Care
Brief Title: Chronic Kidney Disease Clinical Decision Support
Acronym: CKD-CDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: A17-353; 1R18DK118463-01 (NIH)
Record Dates: First submitted 2019-03-25; First posted 2019-03-26 (Actual); Results first posted 2022-12-01 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2021-08

CONDITIONS: Chronic Kidney Diseases; Hypertension; Diabetes
Keywords: Chronic Kidney Disease; CKD; Clinical Decision Support; Diabetes; Hypertension
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hypertension; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Clinic level cluster randomized study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CKD enhanced clinical decision support (CKD-CDS Intervention) (Experimental): Priority Wizard CDS tool is enhanced to incorporate chronic kidney disease(CKD) management. This presents patients and their primary care providers (PCPs) multiple opportunities to consider an evolving array of timely, evidence-based treatment options to improve CKD care. The CDS also provides CV risk factor management like the basic Priority Wizard present in the usual care arm.
  Interventions: Other: CKD enhanced clinical decision support
- Usual Care (No Intervention): A basic Priority Wizard CDS tool for cardiovascular (CV) risk factor management (previously know as the CV Wizard) includes algorithmically derived identification of high CV risk patients and prioritized treatment suggestions for lipids, Blood Pressure (BP), glycemic control, weight, tobacco, and aspirin use based on distance from goal, current medications, labs, allergies, and safety considerations. Has no decision support specific to CKD care.

INTERVENTIONS:
Other: CKD enhanced clinical decision support — The CKD-CDS intervention provides clinical recommendations at any primary care visit for patients with a deficit in any of 5 key elements of CKD care.
  Arms: CKD enhanced clinical decision support (CKD-CDS Intervention)

SUMMARY:
To prevent serious chronic kidney disease (CKD) complications such as end-stage renal disease and cardiovascular events, better strategies are needed to identify, treat, and refer CKD patients seen in primary care clinics. This project expands an existing and successful Web-based clinical decision support (CDS) system to include key elements of CKD care and rigorously assesses the impact of this intervention on quality of CKD care for patients seen in primary care settings, including better recognition of CKD, better management of blood pressure and glucose, and more timely referral to nephrologists when appropriate. This low-cost and highly scalable intervention has high potential to improve CKD care and translate massive public and private sector investments in health informatics into tangible health benefits for large numbers of patients with CKD.

DETAILED DESCRIPTION:
Clinics are randomly allocated 1:1 through a computer-generated program to either control or intervention.

Control Clinics. All control clinics will continue to use the basic Electronic Medical Record (EMR)-linked CDS for cardiovascular (CV) risk factor management. This CDS includes algorithmically derived identification of high CV risk patients and prioritized treatment suggestions for lipids, Blood Pressure (BP), glycemic control, weight, tobacco, and aspirin use based on distance from goal, current medications, labs, allergies, and safety considerations. The basic CDS does not include information specific to CKD care.

Intervention Clinics. The CKD-CDS intervention provides updated clinical recommendations at any primary care visit for patients meeting inclusion and exclusion criteria. This presents patients and their primary care providers (PCPs) multiple opportunities to consider an evolving array of timely, evidence-based treatment options to improve CKD care. The CKD-CDS intervention is rooted in a series of antecedent studies that developed more limited but successful forms of CDS. From an operational point of view, implementing CKD-CDS at intervention clinics requires a series of 4 distinct steps that occur at every encounter:

Step 1: Data exchange and evaluation: The EMR securely exchanges data with the Web Service at every encounter of patients aged 18-75 triggered by BP entry.

Step 2: Recognition of CKD and presence of care deficits: Patients with stage 3-4 CKD are automatically identified by the Web Service and evaluated using algorithms maintained in the Web service for identification of CKD and for the 5 emphasized care gaps (identification of CKD, BP control, glucose control, Angiotensin converting enzyme inhibitor (ACEI)/Angiotensin receptor blocker (ARB) use if appropriate, and nephrology consultation if appropriate). If the patient has a care gap, the rooming staff receives an immediate best practice advisory (BPA) prompt to print CDS materials for the patient and the provider to review and use for shared decision making. Using a sequence of steps successfully implemented in previous studies, the rooming staff will print the materials and give the lay version to the patient to review while waiting for the provider. A professional version is left on the door for the provider to review before entering the exam room. This approach has been well-liked by our providers to help them be prepared and to engage patients in their care needs before the clinician-patient interaction. PCPs can also optionally view an electronic version of the CDS materials. The CDS can be viewed in real time for any patient by clicking on a button programmed in the EMR encounter display.

Step 3: Use of CKD-CDS recommendations as shared decision-making tools: The participating providers and all rooming staff in the intervention clinics will be trained in the use of the PCP (professional) and patient (low-literacy) versions of the CKD-CDS. For this study, the CDS tool will be adapted to emphasize CKD and, for each identified deficit in CKD care, the CKD-CDS will display patient-specific recommendations consistent with then-current national CKD clinical guidelines; for example: (a) recognize CKD and ask the PCP to enter a CKD diagnosis on the problem list if indicated, and/or (b) specific considerations for how to modify BP control, glucose control, or ACEI/ARB therapy, and/or (c) refer certain patients to nephrology when referral criteria are met. The PCP assesses patient preference for any of the CKD-related treatment options. If the patient wants to act on 1 or more, the PCP can address it then or schedule a subsequent visit for that purpose. If the patient is not interested in any option, no further action is needed at that day's visit. The decision support provided to the PCP is very specific and, if pharmacotherapy is indicated, decision support specifies either initiation or titration of specific drugs based on the drugs/doses the patient is currently taking, distance from goal, and other clinical considerations outlined above. The patient version of the CKD-CDS uses symbols to provide easy patient recognition of priority clinical areas and then suggests potential treatment options they can discuss with their provider. Presenting key CKD care recommendations when indicated (all of which are evidence based and capable of improving CKD care) allows the patient freedom to select his or her preferred treatment option from among several potentially beneficial treatment options. Because patient readiness to take health-related actions varies across specific actions, offering several options improves the chance that a given patient may be interested in addressing at least 1 of the evidence-based options presented. Moreover, patient readiness to act is a key predictor of subsequent adherence and success of treatment, as we have previously shown in this patient population. It is important to realize that the printed page the patient receives frames the discussion to a set of prioritized evidence-based treatment options with likely benefit to the patient.

Step 4. Take action based on the decisions made: After discussing with the patient, the provider can then go ahead and order the recommendations suggested by the CDS such as labs, medication, e-consults with nephrology, and referrals to specialists. All actions taken are also based on the provider's clinical judgement.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 75 years, inclusive. The evidence-based guidelines on which the CDS intervention is based are not applicable outside this age range.
2. Have confirmed CKD based on 2 or more estimated glomerular filtration rate (eGFR) values <60 cc/min/1.73m2, including the most recent eGFR value and a previous eGFR at least one week prior
3. Have a CKD care component suboptimally managed as defined by one or more of the following:

   1. Have two or more BP values from separate encounter dates of >=130/80 including the most recent BP to the index visit
   2. Have an individualized A1C over goal as determined by CDS algorithm criteria of most recent glycated hemoglobin (A1C) > 7% OR > 8% if any of the following conditions are identified: cardiovascular disease (CVD) or calculated 10-yr atherosclerotic cardiovascular disease (ASCVD) risk >30%, cancer, hypoglycemia, cognitive impairment, on 2 or more glycemia medications with insulin, or on 3 or more non-insulin glycemia medications
   3. Have most recent eGFR 30-59 with hypertension identified or albumin to creatinine ratio (ACR) > 30 mg/g and not on an ACEI or ARB
   4. Have non-steroidal anti-inflammatory drug (NSAID) other than aspirin on the active medication list
   5. Have a eGFR 15-29 or ACR > 300 mg/g without a nephrology visit in the last 12 months

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from receiving the

CKD-CDS:

1. Patients enrolled in hospice,
2. Patients with active cancer or undergoing chemotherapy
3. Patients with pregnancy in the last year
4. Patients with end stage renal disease

Individuals who meet all inclusion and exclusion criteria at an index visit and have at least one post-index visit in the following 12 months will be included in the primary analyses.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6295 (Actual)
Dates: Start 2019-04-17 (Actual); Primary Completion 2021-09-29 (Actual); Study Completion 2021-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: JoAnn M Sperl-Hillen, MD, Principal Investigator — Senior Investigator, HealthPartners Institute
Locations (1):
- HealthPartners Care System, Bloomington, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] National Kidney Foundation. K/DOQI clinical practice guidelines for chronic kidney disease: evaluation, classification, and stratification. Am J Kidney Dis. 2002 Feb;39(2 Suppl 1):S1-266. No abstract available. PMID 11904577
- [Background] Inker LA, Astor BC, Fox CH, Isakova T, Lash JP, Peralta CA, Kurella Tamura M, Feldman HI. KDOQI US commentary on the 2012 KDIGO clinical practice guideline for the evaluation and management of CKD. Am J Kidney Dis. 2014 May;63(5):713-35. doi: 10.1053/j.ajkd.2014.01.416. Epub 2014 Mar 16. PMID 24647050
- [Background] Stevens PE, Levin A; Kidney Disease: Improving Global Outcomes Chronic Kidney Disease Guideline Development Work Group Members. Evaluation and management of chronic kidney disease: synopsis of the kidney disease: improving global outcomes 2012 clinical practice guideline. Ann Intern Med. 2013 Jun 4;158(11):825-30. doi: 10.7326/0003-4819-158-11-201306040-00007. PMID 23732715
- [Background] Whelton PK, Carey RM, Aronow WS, Casey DE Jr, Collins KJ, Dennison Himmelfarb C, DePalma SM, Gidding S, Jamerson KA, Jones DW, MacLaughlin EJ, Muntner P, Ovbiagele B, Smith SC Jr, Spencer CC, Stafford RS, Taler SJ, Thomas RJ, Williams KA Sr, Williamson JD, Wright JT Jr. 2017 ACC/AHA/AAPA/ABC/ACPM/AGS/APhA/ASH/ASPC/NMA/PCNA Guideline for the Prevention, Detection, Evaluation, and Management of High Blood Pressure in Adults: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. J Am Coll Cardiol. 2018 May 15;71(19):e127-e248. doi: 10.1016/j.jacc.2017.11.006. Epub 2017 Nov 13. No abstract available. PMID 29146535
- [Background] Andrade SE, Gurwitz JH, Field TS, Kelleher M, Majumdar SR, Reed G, Black R. Hypertension management: the care gap between clinical guidelines and clinical practice. Am J Manag Care. 2004 Jul;10(7 Pt 2):481-6. PMID 15298234
- [Background] Grant RW, Cagliero E, Dubey AK, Gildesgame C, Chueh HC, Barry MJ, Singer DE, Nathan DM, Meigs JB. Clinical inertia in the management of Type 2 diabetes metabolic risk factors. Diabet Med. 2004 Feb;21(2):150-5. doi: 10.1111/j.1464-5491.2004.01095.x. PMID 14984450
- [Background] Phillips LS, Ziemer DC, Doyle JP, Barnes CS, Kolm P, Branch WT, Caudle JM, Cook CB, Dunbar VG, El-Kebbi IM, Gallina DL, Hayes RP, Miller CD, Rhee MK, Thompson DM, Watkins C. An endocrinologist-supported intervention aimed at providers improves diabetes management in a primary care site: improving primary care of African Americans with diabetes (IPCAAD) 7. Diabetes Care. 2005 Oct;28(10):2352-60. doi: 10.2337/diacare.28.10.2352. PMID 16186262
- [Background] van Dipten C, van Berkel S, van Gelder VA, Wetzels JFM, Akkermans RP, de Grauw WJC, Biermans MCJ, Scherpbier-de Haan ND, Assendelft WJJ. Adherence to chronic kidney disease guidelines in primary care patients is associated with comorbidity. Fam Pract. 2017 Aug 1;34(4):459-466. doi: 10.1093/fampra/cmx002. PMID 28207923
- [Background] O'Connor PJ, Sperl-Hillen JM, Rush WA, Johnson PE, Amundson GH, Asche SE, Ekstrom HL, Gilmer TP. Impact of electronic health record clinical decision support on diabetes care: a randomized trial. Ann Fam Med. 2011 Jan-Feb;9(1):12-21. doi: 10.1370/afm.1196. PMID 21242556
- [Background] Sperl-Hillen JM, O'Connor PJ, Averbeck BM, et al. Outpatient EHR-based diabetes clinical decision support that works: lessons learned from implementing Diabetes Wizard. Diabetes Spectrum. 2010;23(3):150-154
- [Background] Kharbanda EO, Nordin JD, Sinaiko AR, Ekstrom HL, Stultz JM, Sherwood NE, Fontaine PL, Asche SE, Dehmer SP, Amundson JH, Appana DX, Bergdall AR, Hayes MG, O'Connor PJ. TeenBP: Development and Piloting of an EHR-Linked Clinical Decision Support System to Improve Recognition of Hypertension in Adolescents. EGEMS (Wash DC). 2015 Jul 9;3(2):1142. doi: 10.13063/2327-9214.1142. eCollection 2015. PMID 26290886
- [Background] Gilmer TP, O'Connor PJ, Sperl-Hillen JM, Rush WA, Johnson PE, Amundson GH, Asche SE, Ekstrom HL. Cost-effectiveness of an electronic medical record based clinical decision support system. Health Serv Res. 2012 Dec;47(6):2137-58. doi: 10.1111/j.1475-6773.2012.01427.x. Epub 2012 May 11. PMID 22578085
- [Background] Hargraves I, LeBlanc A, Shah ND, Montori VM. Shared Decision Making: The Need For Patient-Clinician Conversation, Not Just Information. Health Aff (Millwood). 2016 Apr;35(4):627-9. doi: 10.1377/hlthaff.2015.1354. PMID 27044962
- [Background] Agoritsas T, Heen AF, Brandt L, Alonso-Coello P, Kristiansen A, Akl EA, Neumann I, Tikkinen KA, Weijden Tv, Elwyn G, Montori VM, Guyatt GH, Vandvik PO. Decision aids that really promote shared decision making: the pace quickens. BMJ. 2015 Feb 10;350:g7624. doi: 10.1136/bmj.g7624. PMID 25670178
- [Derived] Sperl-Hillen J, Crain AL, Wetmore JB, Chumba LN, O'Connor PJ. A CKD Clinical Decision Support System: A Cluster Randomized Clinical Trial in Primary Care Clinics. Kidney Med. 2023 Dec 12;6(3):100777. doi: 10.1016/j.xkme.2023.100777. eCollection 2024 Mar. PMID 38435072

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Clinics are randomly allocated 1:1 through a computer-generated program to either control or intervention. Patients who have their index visit at a control clinic are assigned to the usual care group and patients who have their index visit at an intervention clinic are assigned to the CKD-CDS intervention group.
Units Other Than Participants: Clinics
Period: Overall Study
Arm/Group | CKD Enhanced Clinical Decision Support (CKD-CDS Intervention) | Usual Care
Started | 2923; 16 Clinics | 3372; 16 Clinics
Completed | 2923; 16 Clinics | 3372; 16 Clinics
Not Completed | 0; 0 Clinics | 0; 0 Clinics

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CKD Enhanced Clinical Decision Support (CKD-CDS Intervention) | Usual Care | Total
Number analyzed (Participants) | 2923 | 3372 | 6295
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1078 | 1254 | 2332
  >=65 years | 1845 | 2118 | 3963
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1602 | 1954 | 3556
  Male | 1321 | 1418 | 2739
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 44 | 77 | 121
  Not Hispanic or Latino | 2838 | 3258 | 6096
  Unknown or Not Reported | 41 | 37 | 78
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 11 | 16 | 27
  Asian | 119 | 142 | 261
  Native Hawaiian or Other Pacific Islander | 3 | 7 | 10
  Black or African American | 274 | 250 | 524
  White | 2439 | 2853 | 5292
  More than one race | 5 | 7 | 12
  Unknown or Not Reported | 72 | 97 | 169
Region of Enrollment [Number; unit: participants]
  United States | 2923 | 3372 | 6295
CKD Diagnosis [Count of Participants; unit: Participants] — Provider-diagnosed CKD among patients with laboratory evidence of stage 3-4 CKD and no prior diagnosis.
  Participants | 1355 | 1589 | 2944

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With CKD Diagnosis
Description: Number of patients who had a CKD diagnosis document in the 18 months post index.
Time Frame: 18-month period post index
Measure: Count of Participants; unit: Participants
Arm/Group | CKD Enhanced Clinical Decision Support (CKD-CDS Intervention) | Usual Care
Number analyzed (Participants) | 1568 | 1783
Participants | 417 | 389
Statistical Analysis 1: Comparison: CKD Enhanced Clinical Decision Support (CKD-CDS Intervention) vs Usual Care; Test type: Superiority; p = .21, Mixed Models Analysis; Risk Ratio (RR) = 1.17, 95% CI 2-sided [.91 to 1.51], Standard Error of Mean 0.12

2. Primary Outcome: Number of Patients With Orders for Angiotensin-converting Enzyme Inhibitors (ACEI) or Angiotension II Reception Blockers (ARB)
Description: Number of patients who had an Angiotensin-converting enzyme inhibitors (ACEI) or Angiotension II reception blockers (ARB) order in the 18 months post index.
Time Frame: 18-month period post index
Measure: Count of Participants; unit: Participants
Arm/Group | CKD Enhanced Clinical Decision Support (CKD-CDS Intervention) | Usual Care
Number analyzed (Participants) | 952 | 1192
Participants | 151 | 192
Statistical Analysis 1: Comparison: CKD Enhanced Clinical Decision Support (CKD-CDS Intervention) vs Usual Care; Test type: Superiority; p = .61, Mixed Models Analysis; Risk Ratio (RR) = .95, 95% CI 2-sided [.76 to 1.18], Standard Error of Mean 0.11

3. Primary Outcome: Number of Patients With Optimal Blood Pressure Control
Description: Number of patients for whom the average of the two most recent blood pressures prior to 18 months post index was <130/80.
Time Frame: 18-month period post index
Measure: Count of Participants; unit: Participants
Arm/Group | CKD Enhanced Clinical Decision Support (CKD-CDS Intervention) | Usual Care
Number analyzed (Participants) | 1633 | 1719
Participants | 334 | 388
Statistical Analysis 1: Comparison: CKD Enhanced Clinical Decision Support (CKD-CDS Intervention) vs Usual Care; Test type: Superiority; p = .84, Mixed Models Analysis; Risk Ratio (RR) = .98, 95% CI 2-sided [0.84 to 1.15], Standard Error of Mean 0.08

4. Primary Outcome: Number of Patients With Optimal Glucose Control
Description: Number of patients whose last A1c was <7% in the 1-18 months post index.
Time Frame: 1 to 18-month period post index
Measure: Count of Participants; unit: Participants
Arm/Group | CKD Enhanced Clinical Decision Support (CKD-CDS Intervention) | Usual Care
Number analyzed (Participants) | 659 | 719
Participants | 141 | 159
Statistical Analysis 1: Comparison: CKD Enhanced Clinical Decision Support (CKD-CDS Intervention) vs Usual Care; Test type: Superiority; p = .99, Mixed Models Analysis; Risk Ratio (RR) = 1.00, 95% CI 2-sided [.8 to 1.24], Standard Error of Mean 0.11

5. Primary Outcome: Number of Patients With Referral to Nephrology
Description: Number of patients who have a referral to nephrology in the 18 months post index.
Time Frame: 18-month period post index
Measure: Count of Participants; unit: Participants
Arm/Group | CKD Enhanced Clinical Decision Support (CKD-CDS Intervention) | Usual Care
Number analyzed (Participants) | 238 | 263
Participants | 92 | 95
Statistical Analysis 1: Comparison: CKD Enhanced Clinical Decision Support (CKD-CDS Intervention) vs Usual Care; Test type: Superiority; p = .86, Mixed Models Analysis; Risk Ratio (RR) = 1.02, 95% CI 2-sided [.79 to 1.32], Standard Error of Mean 0.12

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | CKD Enhanced Clinical Decision Support (CKD-CDS Intervention) | Usual Care
All-Cause Mortality (participants affected / at risk) | 151/2923 | 175/3372
Serious Adverse Events (participants affected / at risk) | 541/2923 | 543/3372
Other Adverse Events (participants affected / at risk) | 1039/2923 | 1100/3372
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CKD Enhanced Clinical Decision Support (CKD-CDS Intervention) (N=2923) | Usual Care (N=3372)
hospitalizations (General disorders) | 541 (2923) | 543 (3372)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | CKD Enhanced Clinical Decision Support (CKD-CDS Intervention) (N=2923) | Usual Care (N=3372)
Emergency Room Visits (General disorders) | 1039 | 1100
hypoglycemia (Endocrine disorders) | 202/1123 | 232/1263
hypotension (Vascular disorders) | 548 | 814
hypokalemia (Metabolism and nutrition disorders) | 853 | 1061
hyperkalemia (Metabolism and nutrition disorders) | 660 | 847

LIMITATIONS AND CAVEATS:
Some Usual Care (UC) participants received CDS for BP and A1c management due to existing CDS pre-dating the study. Due to Corona Virus Disease 2019 (COVID-19), the study paused 5 months, and there were fewer office visits, which would have limited intervention exposure. The intervention didn't allow for video visit screen sharing, a visit type that increased in the pandemic. There was a potential learning effect contamination due to some clinicians caring for patients in both study arms.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-09): https://cdn.clinicaltrials.gov/large-docs/88/NCT03890588/Prot_SAP_000.pdf